CLINICAL TRIAL: NCT06009497
Title: Romiplostim in Combination With Ciclosporin Versus Ciclosporin in the Treatment of Newly Diagnosed Non-severe Aplastic Anemia
Brief Title: Romiplostim in Combination With CsA vs. CsA in the Treatment of Newly Diagnosed NSAA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Romiplostim-1
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Non Severe Aplastic Anemia
MeSH Terms: interventions — romiplostim; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Romiplostim+CsA (Experimental): Romiplostim 10 µg/kg, subcutaneous injection, once a week, for at least 3 months. Patients with platelet count ≥50×109/L can stop using, and continue to use with platelet count < 50×109/L.
  Ciclosporin 3-5mg/kg/d, adjust the dose to keep trough ciclosporin plasma concentration 100-200ng/ml. Ciclosporin should be used for at least 6 months to evaluate the efficacy. Effective patients will continue to use ciclosporin for at least 1.5 years, followed by a slow reduction.
  Interventions: Drug: Romiplostim; Drug: Ciclosporin
- CsA (Experimental): Ciclosporin 3-5mg/kg/d, adjust the dose to keep trough ciclosporin plasma concentration 100-200ng/ml. Ciclosporin should be used for at least 6 months to evaluate the efficacy. Effective patients will continue to use ciclosporin for at least 1.5 years, followed by a slow reduction.
  Interventions: Drug: Ciclosporin

INTERVENTIONS:
Drug: Romiplostim — Romiplostim 10 µg/kg, subcutaneous injection, once a week.
  Arms: Romiplostim+CsA
Drug: Ciclosporin — Ciclosporin 3-5mg/kg/d, adjust the dose to keep trough ciclosporin plasma concentration 100-200ng/ml.

SUMMARY:
Aplastic anemia (AA) is a group of clinical syndromes caused by a significant decrease in bone marrow hematopoietic tissue from different etiologies, resulting in hematopoietic failure. Treatment options for patients with aplastic anemia are very limited. In a phase II/III, multicenter, open-label study exploring the efficacy and safety of romiplostim, the primary endpoint showed an overall response rate of 84% [95% CI 66-95%] at week 27. However, there are no prospective clinical data exploring whether romiplostim combined with ciclosporin (CsA) can further improve efficacy than ciclosporin monotherapy in newly diagnosed NSAA. Therefore, we aimed to compare the efficacy and safety of romiplostim in combination with CsA versus CsA monotherapy.

DETAILED DESCRIPTION:
Aplastic anemia (AA) is a group of clinical syndromes caused by a significant decrease in bone marrow hematopoietic tissue from different etiologies, resulting in hematopoietic failure. Treatment options for patients with aplastic anemia are very limited. By binding to the thrombopoietin (TPO) receptor, thrombopoietin receptor agonists (TPO-RAs) can cause conformational changes in the TPO receptor, activate the JAK2/STATS pathway, and increase megakaryocyte progenitor cells proliferation and platelet production. At present, TPO-RAs including eltrombopag, lusutrombopag, romiplostim, and avatrombopag have been approved by FDA. In a phase II/III, multicenter, open-label study exploring the efficacy and safety of romiplostim, 31 patients with refractory AA were enrolled. The primary endpoint for the proportion of patients who achieved any hematological (platelet, neutrophil, and red blood cell) response at week 27 was 84% [95% CI 66-95%]. At week 53, the three-line response rate was 39% (95% CI 22-58%). However, there are no prospective clinical data exploring whether romiplostim combined with ciclosporin (CsA) can further improve efficacy than ciclosporin monotherapy in newly diagnosed NSAA. Since romiplostim and CsA have good safety, if it is proved that the combination of the two drugs is superior to ciclosporin monotherapy, it can quickly improve blood patterns in NSAA, avoid the use of more expensive ATG, and provide some help to reduce the economic burden of AA patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old.
2. Clearly diagnosed as untreated NSAA.
3. At least one of the following conditions was met at the time of enrollment: hemoglobin <90 g/L. Platelet <30×109/L, neutrophils <1.0×109/L.
4. Baseline liver and kidney function (ALT, AST, Cr) was less than 2 times the normal value.
5. No active infection; Not pregnant or breastfeeding.
6. Agree to sign the consent form.
7. The Eastern Cancer Collaboration Group (ECOG) score was 0-2.

Exclusion Criteria:

1. Pancytopenia caused by other causes, such as myelodysplastic syndrome (MDS).
2. There is cytogenetic evidence of clonal hematologic bone marrow diseases (MDS, AML).
3. PNH clone ≥50%.
4. Had received hematopoietic stem cell transplantation (HSCT) before enrollment.
5. Immunosuppressive therapy such as ATG or cyclosporine use for more than 2 weeks.
6. Infection or bleeding that is not controlled by standard treatment.
7. Allergic to recombinant TPO or Hitrepopar.
8. Active HIV, HCV, HBV infection or cirrhosis, or portal hypertension.
9. Any concomitant malignancy or local basal cell carcinoma of the skin within 5 years.
10. Previous history of thromboembolic events, heart attack or stroke (including antiphospholipid antibody syndrome), and current use of anticoagulants.
11. Women who are pregnant or nursing (lactation).
12. Have participated in other clinical trials within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) | 3, 6 months
  Proportion of patients who achieved complete response and partial response.
complete response rate (CRR) | 3, 6 months
  Proportion of patients who achieved complete response.

SECONDARY OUTCOMES:
adverse event rate | 3, 6 months
  All adverse events that occur or worsen during treatment, as well as those that occur later but are believed by the investigator to be related to the investigational drug, will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young NS. Aplastic anaemia. Lancet. 1995 Jul 22;346(8969):228-32. doi: 10.1016/s0140-6736(95)91273-8. No abstract available. PMID 7616805
- [Background] Young NS. Aplastic Anemia. N Engl J Med. 2018 Oct 25;379(17):1643-1656. doi: 10.1056/NEJMra1413485. No abstract available. PMID 30354958
- [Background] Bacigalupo A. How I treat acquired aplastic anemia. Blood. 2017 Mar 16;129(11):1428-1436. doi: 10.1182/blood-2016-08-693481. Epub 2017 Jan 17. PMID 28096088
- [Background] Yang C, Zhang X. Incidence survey of aplastic anemia in China. Chin Med Sci J. 1991 Dec;6(4):203-7. PMID 1813058
- [Background] Tichelli A, de Latour RP, Passweg J, Knol-Bout C, Socie G, Marsh J, Schrezenmeier H, Hochsmann B, Bacigalupo A, Samarasinghe S, Rovo A, Kulasekararaj A, Roth A, Eikema DJ, Bosman P, Bader P, Risitano A, Dufour C; SAA Working Party of the EBMT. Long-term outcome of a randomized controlled study in patients with newly diagnosed severe aplastic anemia treated with antithymocyte globulin and cyclosporine, with or without granulocyte colony-stimulating factor: a Severe Aplastic Anemia Working Party Trial from the European Group of Blood and Marrow Transplantation. Haematologica. 2020 May;105(5):1223-1231. doi: 10.3324/haematol.2019.222562. Epub 2019 Oct 3. PMID 31582549
- [Background] Kuter DJ. The biology of thrombopoietin and thrombopoietin receptor agonists. Int J Hematol. 2013 Jul;98(1):10-23. doi: 10.1007/s12185-013-1382-0. Epub 2013 Jul 3. PMID 23821332
- [Background] Jing FM, Zhang XL, Meng FL, Liu XM, Shi Y, Qin P, Wang L, Zhou H, Hou Y, Song Q, Peng J, Hou M. Anti-c-Mpl antibodies in immune thrombocytopenia suppress thrombopoiesis and decrease response to rhTPO. Thromb Res. 2018 Oct;170:200-206. doi: 10.1016/j.thromres.2018.08.021. Epub 2018 Aug 30. PMID 30199786
- [Background] Ghanima W, Cooper N, Rodeghiero F, Godeau B, Bussel JB. Thrombopoietin receptor agonists: ten years later. Haematologica. 2019 Jun;104(6):1112-1123. doi: 10.3324/haematol.2018.212845. Epub 2019 May 9. PMID 31073079
- [Background] Jang JH, Tomiyama Y, Miyazaki K, Nagafuji K, Usuki K, Uoshima N, Fujisaki T, Kosugi H, Matsumura I, Sasaki K, Kizaki M, Sawa M, Hidaka M, Kobayashi N, Ichikawa S, Yonemura Y, Enokitani K, Matsuda A, Ozawa K, Mitani K, Lee JW, Nakao S. Efficacy and safety of romiplostim in refractory aplastic anaemia: a Phase II/III, multicentre, open-label study. Br J Haematol. 2021 Jan;192(1):190-199. doi: 10.1111/bjh.17190. Epub 2020 Nov 5. PMID 33152120
- [Background] Ruan J, Zuo W, Chen M, Yang C, Han B. Eltrombopag is effective in patients with relapse/refractory aplastic anemia-report from a single center in China. Ann Hematol. 2020 Dec;99(12):2755-2761. doi: 10.1007/s00277-020-04266-1. Epub 2020 Sep 17. PMID 32944791